CLINICAL TRIAL: NCT06330389
Title: Anesthetic Experience and Patients 'Prognosis of SARS-CoV-2 Positive Versus Negative Burns Patients: An Observational Case -Control Study
Brief Title: Burn Injuries During COVID-19 Pandemic and Its Influence on Length of Stay
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-20-1074
Record Dates: First submitted 2021-08-04; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; burn; outcome; Perioperative; Length of stay
MeSH Terms: conditions — COVID-19; Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Positive and Negative status: Burn injuries with COVID-19 Positive and Negative status underwent surgery
  Interventions: Procedure: Burn Injuries Graft Surgery

INTERVENTIONS:
Procedure: Burn Injuries Graft Surgery — Burn Injuries Graft Surgery

SUMMARY:
Burn injuries were thought to be difficult to treat during the new corona virus epidemic. Our goal is to determine the risk factors that influence length of hospital stay (LOS) of burn injured patients during COVID -19 pandemic.

DETAILED DESCRIPTION:
1. Introduction / History

The world is being attacked by the rapidly expanding severe acute respiratory syndrome coronavirus-2 (SARS-Cov-2) epidemic, which is exacerbating an economic crisis. SARS-Cov-2 is the cause of the coronavirus disease 2019 (COVID-19). Anaesthetists are at risk for contracting a virus while doing their regular duties because they frequently come into touch with respiratory droplets.

All nations have put protective and preventive measures in place, forcing people to spend more time at home. A Brazilian study discovered that during the COVID-19 pandemic period, spending more time at home increased exposure to sanitizing products, which include ethanol and hydrogen peroxides that can cause burn injuries.

Aim of our Study:

Our goal is to determine the risk factors that influence length of hospital stay (LOS) of burn injured patients during COVID -19 pandemic.

Inclusion Criteria:

Patients who had the burn graft surgery at Al Wakrah Hospital; Hamad Medical Corporation between from 1st of April to end of November 2020. Planned number will include all COVID-19 positive and negative subjects in this period.

Data Source The electronic medical record (Cerner) used in order to identify patients who match study defined criteria. The investigators can Collect data directly from Cerner to excel sheet

Variable Abstraction Patient demographic and clinical data will be collected including age, morbidities, presenting symptoms, physical examination, laboratory investigations, intraoperative data, type of surgery, postoperative course, survival, and length of hospital stay and follow up.

In addition, the type of anesthesia is also included as factor for further complications ex general anesthesia, spinal or combined spinal epidural type.

Observation full reviewing of their medical illness and chart laboratory and investigations will be collected after getting approval of MRC and IRB committee.

ELIGIBILITY:
Inclusion Criteria:

* All burn injuries required surgery with COVID-19 positive or negative status

Exclusion Criteria:

* Other surgery during COVID-19 pandemic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had the burn graft surgery at Al Wakrah Hospital; Hamad Medical Corporation between from 1st of April to end of November 2020. Planned number will include all COVID-19 positive and negative.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Our goal is to determine the risk factors that influence length of hospital stay (LOS) of burn injured patients during COVID -19 pandemic. | 60-90 days
  Our goal is to determine the risk factors that influence length of hospital stay (LOS) of burn injured patients during COVID -19 pandemic.

SECONDARY OUTCOMES:
Clinical diffreneces between burn injuries with positive vs negative COVID-19 status | 60-90 days
  Details for those risk Factors: BMI; Pre Op Lab data, Intra Op data ex. blood loss / ml, transfusions/ ml or Unit , surgery time/ min, etc, Post operative data and ICU admission data, , lab parameters, INR,LFTs/unit , required blood transfusions/ml or Unit , re intubation times, vasopressor needs. Analyze lab values /unit, check number of days in hospital stay and ICU stay .
  Analyze risk factors which affect hospital length of stay. Analyze risk factors using cox regression and investigate hazard ratio for each one to determine which is independent risk factor OR associated factor.

CONTACTS AND LOCATIONS:
Locations (1):
- HAMAD Medical Corporation- Al Wakra Hospital, Doha, Qatar

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT06330389/Prot_SAP_000.pdf